CLINICAL TRIAL: NCT04425200
Title: Prevalence of HRR-related Genes Mutations and Prognosis in Metastatic Castration Resistant Prostate Cancer (mCRPC) Patients in Real World Setting
Acronym: ZENSHIN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D081LR00002
Record Dates: First submitted 2020-05-21; First posted 2020-06-11 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Prostatic Neoplasms
Keywords: metastatic castration resistant prostate cancer, BRCA1, BRCA2, ATM, Homologous recombination repair
MeSH Terms: conditions — Prostatic Neoplasms; Fanconi Anemia, Complementation Group D1; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An archived formalin fixed paraffin embedded (FFPE) sample, ten slides and 10 μm in thickness on uncharged slide be used for HRR-related gene mutation testing in principle. And also, ten 10 μm slides is sent to Myriad with one 3-5 micron on a charge slide for the HE staining(Hematoxylin and eosin staining) which is continuous with the slice for HRR-related gene mutation. These contents include with a sample of >25 mm2 in section area containing a ≥30% tumor nuclei preferred (≥20% tumor nuclei accepted). If patients have some tumor samples at multiple points, the latest sample is preferred to use HRR-related gene mutation testing. And other tumor sample is acceptable to use HRR-related gene mutation testing if test is failed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the prevalence of tissue homologous recombination repair (HRR)-related gene mutations (positive/negative/Variant of uncertain significance (VUS)), clinical outcome such as prostate-specific antigen-progression free survival (PSA-PFS), overall survivals (OS) and treatment pattern in mCRPC patients.

<Methods> Study design: multi-center, prospective cohort study

Data Source(s):

In this study, 155 patients (expected recruitment patients: maximum 205 patients) will be enrolled from approximately 20~30 sites in Japan. Study Population: mCRPC patients who diagnosed between 2014 and 2018. Exposure(s): N.A Outcome(s): Prevalence of tissue HRR-related gene mutations, clinical outcomes such as Over survival and PSA-PFS, Treatment pattern

Sample Size Estimations:

The target population is 155 patients based on the prevalence of HRR-related genes (BRCA1, BRCA2 and ATM) which is reported in previous global study (PROfound study).

Statistical Analysis:

This study is not intended to verify specific hypotheses, and the results are evaluated descriptively. There is no plan of interim analyses before the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20, Japanese men at the time of informed consent.
* Patients who provided informed consent. If the patient has died, opt-out will be applicable.
* Patients who are diagnosed as mCRPC between January 1st in 2014 and December 31st in 2018.
* Patients who have a FFPE tumor sample (primary or metastatic) with Formalin Neutral Buffer Solution.
* Patients which the investigator judges to secure the enough amount of tumor samples for future laboratory test.

Exclusion Criteria:

* Patients who have failed HRR-related gene mutation testing with the myChoice HRD plus in screening period.
* Patients who have an only FFPE primary tumor sample (primary or metastatic) with unbuffered formalin including acidic formalin.
* Patients who have taken an investigational medical product for prostate cancer from Jan 1st , 2014 to Dec 31st 2020.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The target population is mCRPC patients who diagnosed between 2014 and 2018 and be confirmed to be succeeded HRR-related gene mutation analysis with archived primary or metastatic tumor sample. As median of expected overall survival of mCRPC is 2.5 to 3 years from diagnosis, follow up period is enough to measure outcomes including survival. The baseline period is set to calculate overall survival and to detect clinical outcome at least half. The patients will be enrolled consecutively to this study.
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of tissue HRR-related gene mutations | Baseline
  Calculate number and prevalence of each HRR-related gene mutation status (Positive/Negative/VUS), respectively. Prevalence will be accompanied by 95% Clopper-Pearson confidence intervals.

SECONDARY OUTCOMES:
Proportion of each treatment pattern | From index date(diagnosed as mCRPC) patients to December 31 2020
  The number (%) of patients by treatment pattern in 1st line treatment, 2nd line, and 3rd line treatment after diagnosed as mCRPC, respectively, will be calculated.

OTHER OUTCOMES:
Patient's characteristics including stratified by tissue HRR-related gene mutations in mCRPC patients | Baseline
  Patient's characteristics will be summarized.
PSA50 response | From index date(diagnosed as mCRPC) to december 31 2020
  PSA50 response will be analysed based on baseline and nadir PSA value in each treatment.

CONTACTS AND LOCATIONS:
Locations (26):
- Japan (26):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Jikei University Kashiwa Hospital, Kashiwa, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Hakodate Goryoukaku Hospital, Hakodate, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagawa University Hospital, Hiragi, Kagawa-ken
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Nara Medical University Hospital, Kashihara, Nara
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Medical Center, Kawagoe, Saitama
  - Tottori University Hospital, Yonago, Tottori
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Chiba University Hospital, Chiba
  - Gifu University Hospital, Gifu
  - Kyoto Prefectural University of Medicine, Kyoto
  - University of Miyazaki Hospital, Miyazaki
  - Okayama University Hospital, Okayama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials/studies via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081LR00002&attachmentIdentifier=af31e80d-5dae-46e5-accb-47980c519713&fileName=SYNOPSIS_for_Clin.govZENSHIN_20211112.pdf&versionIdentifier=